CLINICAL TRIAL: NCT04642235
Title: Nature and Well-Being Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American Heart Association (Other); Pennsylvania Horticultural Society (Unknown); United States Forest Service (Unknown); OLIN Studio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 842575
Record Dates: First submitted 2020-11-13; First posted 2020-11-24 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Environmental Exposure; Health Behavior; Health, Subjective
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nature Nook (Experimental): Nature Nook builds on our prior work with a standard vacant lot greening intervention involving: removing trash, grading the land, planting new grass and trees, installing a low wooden perimeter fence, and regular maintenance. This greening intervention was designed as a blight removal strategy. People in this arm receive no intervention.
  Interventions: Other: Nature Nook
- Nature Coach (Experimental): The Nature Coach intervention, developed in a prior study (NCT04146025), will be delivered to people in their homes. Participants will live in the blocks immediately surrounding the study vacant lots randomized to this arm. The lots in this arm receive no intervention.
  Interventions: Behavioral: Nature Coach
- Nature Nook + Nature Coach (Experimental): This is a combined arm: a place-based intervention (Nature Nook) and a person-based intervention (Nature Coach).
  Interventions: Other: Nature Nook + Nature Coach
- Control (No Intervention): The study lots randomly selected for this arm, as well as the participants living near them, receive no intervention.

INTERVENTIONS:
Other: Nature Nook — The Nature Nook intervention will take place on lots that already have the standard greening intervention. In addition, design elements will be added such as a simple path and benches to explicitly invite people into the space. An additional difference is the exclusive use of larger, corner lots, rather than smaller mid-block spaces, to maximize visibility.
  Arms: Nature Nook
Behavioral: Nature Coach — The Nature Coach Intervention consists of 3 components - home visit, text message follow up, and goal feedback.
  Home visit. During the 1-hour home visit, the coach will (a) provide education about the health benefits of nature, (b) identify nearby nature targets for the participant to visit, (c) complete a pre-commitment contract based on individualized weekly nature goals, and (d) brainstorm barriers and solutions to reaching the goals.
  Personalized weekly text messages. Texts will serve as reminders of goals set with the Nature Coach, as well as encouragement to meet the goals. The context of text messages with change slightly based on individual participants, the goals they set, and the barriers they identify.
  Goal feedback- At the end of each week, participants will receive a progression badge via text message that shows the amount of days and time they spent in nature, and how this matched up to the goal set with the Nature Coach.
  Arms: Nature Coach
Other: Nature Nook + Nature Coach — The combined intervention will involve the installation of Nature Nooks to blighted vacant lots followed by the delivery of the Nature Coach intervention to people living in the immediate surrounding blocks. The intervention will be tailored to explicitly direct participants to use the Nature Nook.
  Arms: Nature Nook + Nature Coach

SUMMARY:
The investigators pilot test two intervention strategies to increase green space use- place-based and person-based, as well as evaluate the dose-response relationship between green space use and health.

DETAILED DESCRIPTION:
Neighborhood conditions can positively impact mental health and wellbeing. Green space has been cited as a potential buffer between inequitable neighborhood conditions and poor health. However, there is limited evidence how to increase exposure to green space and how much exposure is needed to produce benefit. Place-based and person-based interventions offer contrasting approaches to improving the impact of the environment on health. The environment influences people as they traverse the spaces between home, work, and recreation, in ways that can be healthy or harmful. Place-based approaches directly change the environment to encourage healthy behaviors, and potentially have broad population impact. Alternatively, person-based approaches directly target individuals' behavior and may be more feasible. To our knowledge, no studies combine both approaches into a single intervention, which may be more effective over either alone.

The broad objectives of this proposal are to pilot test two intervention strategies to increase green space use- place-based and person-based, as well as evaluate the dose-response relationship between green space use and health. Our place-based intervention, Nature Nooks, builds on our prior greening treatment by adding new features to encourage use - a path and benches to invite people into the space and instillation on large corner lots to maximize visibility. The investigators develop our person-based intervention, Nature Coach, as a novel adoption of an analogous, established patient navigator concept in healthcare.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Live in one of the 8 target neighborhoods identified
* Have a smartphone
* Able to understand and respond to an oral interview in English.

Exclusion Criteria:

* Unwilling to go outside
* Not ambulatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Green Space Use | 12 months
  This will measured using GPS data to see the amount of time spent in green space.

SECONDARY OUTCOMES:
Mental health and well-being: CES-D | 12 months
  This will be measured using the Center for Epidemiologic Studies - Depression Scale (CES-D). The CES-D scale is a brief 20-item self-report scale designed to measure self-reported symptoms associated with depression experienced in the past week. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms. A score of 16 points or more is considered depressed.
Mental health and well-being: PSS-10 | 12 months
  The Perceived Stress Scale-10(PSS-10) is a self-report instrument consisting of 10 items to assess stress perception, with the time frame being during the last month. Each of the items on the PSS-10 are rated on a 5-point Likert scale (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often). Four positively stated items (item 4, 5, 7, and 8) are reversely scored (0 = very often, 1 = fairy often, 2 = sometimes, 3 = almost never, 4 = never). The sum of the 10 items represents the total score, with higher scores representing higher levels of perceived stress.
Mental health and well-being: WHO-5 | 12 months
  The WHO-5 Well-Being Index is a questionnaire that measures current mental well-being, with the time frame being the previous two weeks. This is five items rated on 6-point Likert scale (All of the time, Most of the time, More than half the time, Less than half the time, Some of the time, At no time). The raw score is calculated by totaling the figures of the five answers. The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia South, MD MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Department of Emergency Medicine, Philadelphia, Pennsylvania, United States